CLINICAL TRIAL: NCT02831517
Title: A Phase 1 Pharmacokinetics and Safety Study of BIIB074 in Healthy Japanese and Caucasian Subjects
Brief Title: PK and Safety Study of BIIB074 in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 802HV106; 2016-000874-39 (EudraCT Number)
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Healthy; Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): 48 participants: Cohorts 1,2 and 3 (Single Ascending Dose of BIIB074 or placebo) in a 6:2 ratio
  Interventions: Drug: BIIB074; Drug: Placebo
- Part 2 (Experimental): 16 participants: Multiple Ascending Dosing of BIIB074 or placebo in a 6:2 ratio; 3 times daily [TID] in cohort 4 for 6 days and one time (QD) for 1 day and 2 times daily [BID] in cohort 5 for 6 days and QD for 1 day
  Interventions: Drug: BIIB074; Drug: Placebo

INTERVENTIONS:
Drug: BIIB074 — Administered as specified in the treatment arm
  Other Names: CNV1014802
Drug: Placebo — Matched Placebo

SUMMARY:
The primary objectives of this study are: To evaluate pharmacokinetics (PK) properties of BIIB074 administered as a single oral dose in healthy Japanese and Caucasian participants; and To evaluate the PK properties of BIIB074 administered as repeated oral doses in healthy Japanese participants. The secondary objective of this study is to assess the safety and tolerability of BIIB074 administered as a single oral dose (Japanese and Caucasian participants) and as repeated oral doses (Japanese participants).

ELIGIBILITY:
Key Inclusion Criteria:

* Japanese or Caucasian.
* Japanese participants must have been born in Japan, and their biological parents and grandparents must all have been of Japanese origin.
* Must have a body mass index between 18 and 30 kg/m2, inclusive.

Key Exclusion Criteria:

* Previous exposure to BIIB074, with the exception that Japanese participants who complete Part 1.
* Use of any oral, injected, or implanted hormonal method of contraception that contains ethinyl estradiol within 28 days of Day -1 and an unwillingness to refrain from product use during study participation.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Part 1: PK of BIIB074 single oral dose as assessed by maximum observed concentration (Cmax ) | 15 minutes prior to dosing up to 96 hours post dose
Part 1: PK of BIIB074 single oral dose as assessed by time to reach Cmax (tmax) | 15 minutes prior to dosing up to 96 hours post dose
Part 1: PK of BIIB074 single oral dose as assessed by area under the concentration time curve from time 0 extrapolated to infinity (AUCinf) | 15 minutes prior to dosing up to 96 hours post dose
Part 1: PK of BIIB074 single oral dose as assessed by area under the concentration time curve from time 0 to time of the last measurable drug concentration (AUC0-t) | 15 minutes prior to dosing up to 96 hours post dose
Part 1: PK of BIIB074 single oral dose as assessed by terminal elimination half-life (t1/2) | 15 minutes prior to dosing up to 96 hours post dose
Part 1: PK of BIIB074 single oral dose as assessed by apparent volume of distribution (Vd/F) | 15 minutes prior to dosing up to 96 hours post dose
Part 1: PK of BIIB074 single oral dose as assessed by apparent total body clearance (CL/F) | 15 minutes prior to dosing up to 96 hours post dose
Part 1: PK of BIIB074 single oral dose as assessed by metabolite to parent ratio in AUC (MRAUC) | 15 minutes prior to dosing up to 96 hours post dose
Part 2: PK of BIIB074 repeated oral dose as assessed by Cmax | 15 minutes prior to dosing on Day 1 up to 96 hours post dose on Day 7
Part 2: PK of BIIB074 repeated oral dose as assessed by tmax | 15 minutes prior to dosing on Day 1 up to 96 hours post dose on Day 7
Part 2: PK of BIIB074 repeated oral dose as assessed by area under the concentration time curve within a dosing interval (AUCtau) | 15 minutes prior to dosing on Day 1 up to 96 hours post dose on Day 7
Part 2: PK of BIIB074 repeated oral dose as assessed by trough concentration after repeated doses (Ctrough) | 15 minutes prior to dosing on Day 1 up to 96 hours post dose on Day 7
Part 2: PK of BIIB074 repeated oral dose as assessed by t1/2 | 15 minutes prior to dosing on Day 1 up to 96 hours post dose on Day 7
Part 2: PK of BIIB074 repeated oral dose as assessed by apparent volume of distribution at steady state (Vss/F) | 15 minutes prior to dosing on Day 1 up to 96 hours post dose on Day 7
Part 2: PK of BIIB074 repeated oral dose as assessed by apparent clearance at steady state (CLss/F) | 15 minutes prior to dosing on Day 1 up to 96 hours post dose on Day 7
Part 2: PK of BIIB074 repeated oral dose as assessed by accumulation ratio (Rac) | 15 minutes prior to dosing on Day 1 up to 96 hours post dose on Day 7
Part 2: PK of BIIB074 repeated oral dose as assessed by MRAUC | 15 minutes prior to dosing on Day 1 up to 96 hours post dose on Day 7

SECONDARY OUTCOMES:
Number of participants experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 2 weeks post Part 2 of the Treatment Period
Number of participants with clinically significant laboratory assessment abnormalities | Up to 2 weeks post Part 2 of the Treatment Period
Number of participants with clinically significant vital sign abnormalities | Up to 2 weeks post Part 2 of the Treatment Period
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | Up to 2 weeks post Part 2 of the Treatment Period
Number of participants with clinically significant physical examinations abnormalities | Up to 2 weeks post Part 2 of the Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Leeds, United Kingdom